CLINICAL TRIAL: NCT06812728
Title: Neoadjuvant FOLFIRINOX and Preoperative Chemoradiotherapy Versus Standard Total Neoadjuvant Approach for Locally Advanced Rectal Cancer Patients: a Randomized Controlled Phase 2 Trial.
Brief Title: Neoadjuvant FOLFIRINOX and Preoperative Chemoradiotherapy for Locally Advanced Rectal Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, yostena nagy kamel mekhail, Primary Investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R2025
Record Dates: First submitted 2025-02-01; First posted 2025-02-06 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Rectum Cancer
Keywords: Neoadjuvant; mFOLFIRINOX; TNT; Watch and wait approach; Complete clinical response; Sphincter sparing
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (mFolfox6) (Active Comparator): Chemotherapy (mFolfox6) then radiochemotherapy
  Interventions: Drug: mFolfox6
- Arm B (mFOLFIRINOX) (Experimental): Chemotherapy (mFOLFIRINOX) then radiochemotherapy
  Interventions: Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: mFOLFIRINOX — Neoadjuvant chemotherapy
  Arms: Arm B (mFOLFIRINOX)
Drug: mFolfox6 — Neoadjuvant chemotherapy
  Arms: Arm A (mFolfox6)

SUMMARY:
A phase II clinical trial compared standard TNT (mFolfox6 and CRT) with preoperative chemoradiotherapy (CRT) with neoadjuvant chemotherapy (CT) containing mFolfirinox in patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
This open-label randomized, two-arm phase II trial compared the standard total neoadjuvant approach (TNT) with neoadjuvant CT with mFolfirinox and preoperative CRT in patients with locally advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven rectal adenocarcinoma.
2. Stages cT3 with risk of local recurrence, cT4, or N positive, M0 and for which a multidisciplinary meeting recommend TNT.
3. Resectable tumor, or considered as potentially resectable after CRT.
4. No distant metastases.
5. Patient eligible for surgery
6. World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) performance status 0/1.
7. No heart failure or coronary heart disease symptoms (even controlled).
8. No peripheral neuropathy > grade 1.
9. No prior radiotherapy of the pelvis for any reason and no previous CT
10. No major comorbidity that may preclude the delivery of treatment
11. Adequate contraception in fertile patients.
12. Adequate hematologic function.

13 Adequate hepatic function.

14. Signed written informed consent.

Exclusion Criteria:

1. Metastatic disease
2. Unresectable rectal cancer, including prostatic involvement or extension to pelvic floor muscles Contraindication to 5-FU, or to oxaliplatin or to irinotecan, including Gilbert disease or genotype UGT1A1
3. Medical history of chronic diarrhea or inflammatory disease of the colon or rectum
4. Medical history of angina pectoris or myocardial infarction
5. Other concomitant cancer.
6. Pregnant or breast-feeding woman.
7. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol or follow-up schedule.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2027-01-25 (Estimated); Study Completion 2027-02-25 (Estimated)

PRIMARY OUTCOMES:
Complete clinical response rate | 6 months
  an absence of clinical, endoscopic or imaging evidence of a rectal tumor during the restaging of a patient with locally advanced rectal cancer after neoadjuvant therapy.

SECONDARY OUTCOMES:
Toxicity of chemotherapy | 6 months
  Common Terminology Criteria for Adverse Events (CTCAE) v 5
complete pathological response rectal cancer | 6 months
  the absence of malignant cells on the specimen of rectal resection in patients who were previously treated with neoadjuvant CRT.
disease-free survival | 3 years
  Disease-free survival (DFS) will be defined as the time from randomization to recurrence of tumor or death
Overall survival | 5 years
  Overall survival will be defined as the time from randomisation to the time of occurrence of the first death regardless to its cause. Patients alive at the time of analysis will be censored at the date of the last follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Yostena Mekhail, MD,PhD, Principal Investigator — Menoufia University
Locations (1):
- Medicine, Shibīn al Kawm, Menoufia, Egypt